CLINICAL TRIAL: NCT06297096
Title: Multicentre Clinical Trial Evaluating the Safety and Efficacy of the Combination of Nintedanib+Tocilizumab Compared to Standard Treatment in Patients With Systemic Sclerosis and Interstitial Lung Disease. Analysis With Theranostic Approach
Brief Title: Study of the Efficacy of Nintedanib+Tocilizumab in Patients With Systemic Sclerosis and Interstitial Lung Disease
Acronym: NINTOC-TU
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIGRIR_004NINTOC-TU
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Systemic Sclerosis; Interstitial Lung Disease
Keywords: systemic sclerosis; ILD; tocilizumab; nintedanib; combination therapy
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial | interventions — tocilizumab; nintedanib; Standard of Care; Mycophenolic Acid; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined therapy Nintedanib + Tocilizumab with or without standard treatment + extended diagnostics (Experimental): tocilizumab pre-filled syringe 162 mg subcutaneously once a week nintedanib tablets 150 mg twice a day or 2 x 100 mg a day
  Interventions: Drug: Tocilizumab; Drug: Nintedanib; Drug: Standard therapy
- standard treatment (reference group) + extended diagnostics (Active Comparator): mycophenolate mofetil stable dose from 1000 - 3000 mg daily tablet 500 mg or 250 mg regardless of the preparation (Mycofit, CellCept, Mycophenolate mofetil, Myfenax) or methotrexate 10-25 mg/week orally or subcutaneously as above, regardless of the preparation
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 162 mg s.c./week
  Arms: combined therapy Nintedanib + Tocilizumab with or without standard treatment + extended diagnostics
Drug: Nintedanib — Nintedanib - established doses of nintedanib for adults in the treatment of ILD, also SSc-ILD: 2 x 150 mg daily, in the event of e.g. increased liver enzyme levels, poorer treatment tolerance (e.g. diarrhea), the dose can be reduced to 2 x 100 mg
  Arms: combined therapy Nintedanib + Tocilizumab with or without standard treatment + extended diagnostics
Drug: Standard therapy — mycophenolate mofetil stable dose from 1000 - 3000 mg daily tablet 500 mg or 250 mg regardless of the preparation (Mycofit, CellCept, Mycophenolate mofetil, Myfenax) or methotrexate 10-25 mg/week orally or subcutaneously as above, regardless of the preparation
  Other Names: mycophenolate mofetil; methotrexate

SUMMARY:
The study includes adult patients with systemic sclerosis (SSc) with interstitial lung disease (ILD) to evaluate the efficacy and safety of nintedanib plus tocilizumab combination therapy compared to standard therapy (methotrexate, mycophenolate mofetil) for 56 weeks.

DETAILED DESCRIPTION:
Full title of the trial:

A multicentre clinical trial evaluating the safety and efficacy of the combination of nintedanib and tocilizumab compared to standard treatment in patients with systemic sclerosis and interstitial lung disease. Analysis with theranostic approach and assessment of cytokine activity, markers of inflammation and pulmonary fibrosis using computed tomography, positron emission tomography, and metabolome and transcriptome studies in selected patients. NINTOC-TU study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-74 at the date of signing the informed consent.
2. Written informed consent in accordance with the International Harmonization Guidelines Harmonized Tripartite: Guidelines for Good Clinical Practice (ICH-GCP) and local regulations signed before any study procedure.
3. Documented diagnosis of systemic sclerosis according to the criteria of the American College of Rheumatology (ACR) and The European Alliance of Associations for Rheumatology (former name - European League Against Rheumatism) - EULAR, meeting the criteria of active disease [patients with limited and diffused SSc)] and with an overall disease duration of less than or equal to (≤ 72 months).
4. Patients with interstitial lung disease (ILD) confirmed by HRCT (min. 10% lung involvement).
5. Evaluation of skin induration with the modified Rodnan skin score (mRSS) from 10 to 45 units inclusive.
6. Patients treated with conventional drugs such as mycophenolate mofetil, methotrexate; should be on stable doses for ≥ 8 weeks before and including the screening visit (W0).
7. Patients may be treated with standard therapy, but no new therapy or withdrawal of therapy within 8 weeks before the first screening visit (W0).
8. Patients taking oral glucocorticosteroids (GCS) should be on a stable dose of ≤ 10 mg/day prednisone or equivalent for at least 8 weeks before the baseline visit.
9. Patients of childbearing potential should agree to abstain from sexual activity or use a highly effective method of contraception throughout the study and for at least 3 months after the last dose of medicinal products.

Exclusion Criteria:

1. Patients not fully capable of giving informed consent.
2. Pregnant or breastfeeding women.
3. Major surgery within 8 weeks before screening (W0A).
4. Rheumatic disease other than systemic sclerosis (systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease). Diagnosis of secondary Sjögren's syndrome is acceptable.
5. Active diverticulitis and severe enteritis.
6. Untreated lipid disorders (Initiation of treatment and modification of the lipid profile enable re-screening for examination after 8 weeks from the start of hypolipidemic treatment).
7. Immunization with a live or attenuated vaccine within 4 weeks before scheduled treatment.
8. Known hypersensitivity to human, humanized or murine monoclonal antibodies and hypersensitivity to peanut, soya.
9. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels greater than 1.5 times the upper limit of normal (ULN). If normalized, the patient may be considered for re-screening.
10. Bilirubin >1.5 x ULN.
11. Creatinine clearance <30 ml/min.
12. Significant pulmonary hypertension (PH).
13. Airway obstruction (forced expiratory volume before bronchodilation in 1 second (FEV1)/FVC <0.7) and other clinically significant pulmonary abnormalities.
14. Cardiovascular diseases with heart failure NYHA III/IV.
15. More than 4 digital ulcers or a history of severe digital necrosis requiring hospitalization or severe other digital ulcers.
16. Bleeding risk (such as bleeding tendency, fibrinolysis, full dose of anticoagulants, high dose of antiplatelet therapy, history of central nervous system (CNS) bleeding events in the last year. (INR) >2, prothrombin time (PT) and partial thromboplastin (PTT) > 1.5 x ULN) and history of a thrombotic event within the last year, history of thrombosis still requiring full therapeutic anticoagulant therapy, fibrinolysis or high-dose antiplatelet therapy > 150 mg ASA per day.
17. History of stroke, or myocardial infarction within 6 months before screening.
18. Prior treatment with pirfenidone or nintedanib if a minimum of 6 months had not been completed before enrolling the patient in the NINTOC-TU study.
19. Plasmapheresis and/or plasma exchange within the last 12 weeks before screening and use of immunoglobulins within the last 12 weeks and treatment with tocilizumab, treatments targeting B cell depletion, biologics (e.g. tumor necrosis factor antagonists), tyrosine kinase inhibitors, current treatment with alkylating agents (chlorambucil), autologous bone marrow transplantation, thalidomide, antithymocyte globulin, extracorporeal photopheresis.
20. Treatment with prednisone >10 mg/day, azathioprine, hydroxychloroquine, colchicine, D-penicillamine, sulfasalazine if within 8 weeks before W0. Cyclophosphamide within < 8 weeks of randomization visit (W 1). Rituximab within 6 months of visit (randomization W1).
21. Unstable (fluctuating) background therapy with mycophenolate mofetil or methotrexate in the last 8 weeks.
22. Patients with chronic liver disease (Child-Pugh A, B, C hepatic impairment).
23. Active or significant history of infection, including treatment with intravenous antibiotics within the last 4 weeks or oral antibiotics within 2 weeks before screening. Including active confirmed tuberculosis or latent tuberculosis without chemoprophylaxis following applicable local recommendations. Active infection with HBV, HCV, Herpes-Zoster virus in the last 12 months. Human Immunodeficiency Virus (HIV) infection.
24. A positive result of the SARS-CoV-2 PCR test during the "0" visit is an exclusion criterion, while a history of infection more than 4 weeks before the screening tests and confirmed by a negative SARS-CoV-2 PCR test is not an exclusion criterion.
25. Active or history of malignancy, except for excised/cured local basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ.
26. Active or past drug or alcohol abuse.
27. The inability to understand and comply with the requirements of the protocol (lack of compliance) excludes from participation in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
The decrease in forced vital capacity (FVC) of the lungs | 56 weeks
  The decrease in forced vital capacity (FVC) of the lungs expressed in ml calculated after 56 weeks of treatment

SECONDARY OUTCOMES:
Change in percent lung involvement | 56 weeks
  Change in percent lung involvement assessed by computed tomography (HRCT%) from baseline to assessment in 56 weeks of study
Assessment of absolute changes in DLCO | 56 weeks
  Assessment of absolute changes in DLCO at week 56 compared to baseline (baseline)
Assessment of the absolute changes in predicted FVC% | 56 weeks
  Assessment of the the absolute changes in predicted FVC% at week 56 from baseline
Change in the Six-minute walk test (6MWT) result | 56 weeks
  Change in the Six-minute walk test (6MWT) result at week 56 compared to the baseline value
Change in the Health Assessment Questionnaire-Disability Index (HAQ-DI) score | 56 weeks
  Change in the Health Assessment Questionnaire-Disability Index (HAQ-DI) score at week 56 (from min. 0 to max.3). Scores of 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability.
A change in the patient's global assessment of disease activity | 56 weeks
  A change in the patient's global assessment of disease activity (Patient's Global Assessment - PtGA), assessment at week 56 - PtGA scoring on Visual Analog Scale from optimal condition - 0 mm (min) to 100 mm (max) - the worse condition.
A change in the physician's global assessment of disease activity | 56 weeks
  A change in the physician's global assessment of disease activity (Physician's Global Assessment - PGA), assessment at week 56 - PGA scoring on Visual Analog Scale from optimal condition - 0 mm (min) to 100 mm (max) - the worse condition.
Assessment of the absolute changes from baseline in total scores in St. George's Respiratory Questionnaire (SGRQ) | 56 weeks
  Assessment of the absolute changes from baseline in total scores in St. George's Respiratory Questionnaire (SGRQ) at 56 weeks. St. George's Respiratory Questionnaire (SGRQ) ranges from 1 to 100, where 0 indicates best health and 100 indicates worst health.
Assessment of absolute changes compared to baseline values on the modified Rodnan skin Score (mRSS) | 56 weeks
  Assessment of absolute changes compared to baseline values on the modified Rodnan skin Score (mRSS) at week 56. mRSS is a semiquantitative score, ranging from 0 (normal) to 3 (severe), used to evaluate the skin thickness in 17 different cutaneous sites (for a total score from 0 (good) to 51 (the worst condition).
Percentage of participants with threshold improvement from baseline in modified Rodnan skin Score (mRSS) | 56 weeks
  Percentage of participants with threshold improvement from baseline in modified Rodnan skin Score (mRSS) at week 56. mRSS is a semiquantitative score, ranging from 0 (normal) to 3 (severe), used to evaluate the skin thickness in 17 different cutaneous sites (for a total score from 0 (good) to 51 (the worst condition).
Percentage of participants with modified Rodnan skin Score (mRSS) improvement greater than or equal to (>/=) 20%, 40%, or 60% | Time frame: from baseline to week 56
  Percentage of participants with modified Rodnan skin Score (mRSS) improvement greater than or equal to (>/=) 20%, 40%, or 60% [time frame: baseline to week 56]. mRSS is a semiquantitative score, ranging from 0 (normal) to 3 (severe), used to evaluate the skin thickness in 17 different cutaneous sites (for a total score from 0 (good) to 51 (the worst condition).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Maślińska, PhD, MD, Principal Investigator — National Institute of Geriatrics,Rheumatology and Rehabilitation
Locations (1):
- Centrum Wsparcia Badań Klinicznych, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richeldi L, Cottin V, Flaherty KR, Kolb M, Inoue Y, Raghu G, Taniguchi H, Hansell DM, Nicholson AG, Le Maulf F, Stowasser S, Collard HR. Design of the INPULSIS trials: two phase 3 trials of nintedanib in patients with idiopathic pulmonary fibrosis. Respir Med. 2014 Jul;108(7):1023-30. doi: 10.1016/j.rmed.2014.04.011. Epub 2014 Apr 29. PMID 24834811
- [Background] Inoue Y, Suda T, Kitamura H, Okamoto M, Azuma A, Inase N, Kuwana M, Makino S, Nishioka Y, Ogura T, Takizawa A, Ugai H, Stowasser S, Schlenker-Herceg R, Takeuchi T. Efficacy and safety of nintedanib in Japanese patients with progressive fibrosing interstitial lung diseases: Subgroup analysis of the randomised, double-blind, placebo-controlled, phase 3 INBUILD trial. Respir Med. 2021 Oct;187:106574. doi: 10.1016/j.rmed.2021.106574. Epub 2021 Aug 12. PMID 34564020
- [Background] Cottin V, Richeldi L, Rosas I, Otaola M, Song JW, Tomassetti S, Wijsenbeek M, Schmitz M, Coeck C, Stowasser S, Schlenker-Herceg R, Kolb M; INBUILD Trial Investigators. Nintedanib and immunomodulatory therapies in progressive fibrosing interstitial lung diseases. Respir Res. 2021 Mar 16;22(1):84. doi: 10.1186/s12931-021-01668-1. PMID 33726766
- [Background] Shima Y, Kawaguchi Y, Kuwana M. Add-on tocilizumab versus conventional treatment for systemic sclerosis, and cytokine analysis to identify an endotype to tocilizumab therapy. Mod Rheumatol. 2019 Jan;29(1):134-139. doi: 10.1080/14397595.2018.1452178. Epub 2018 Apr 9. PMID 29529897
- [Background] Denton CP, De Lorenzis E, Roblin E, Goldman N, Alcacer-Pitarch B, Blamont E, Buch M, Carulli M, Cotton C, Del Galdo F, Derrett-Smith E, Douglas K, Farrington S, Fligelstone K, Gompels L, Griffiths B, Herrick A, Hughes M, Pain C, Pantano G, Pauling J, Prabu A, O'Donoghue N, Renzoni E, Royle J, Samaranayaka M, Spierings J, Tynan A, Warburton L, Ong V. Management of systemic sclerosis: British Society for Rheumatology guideline scope. Rheumatol Adv Pract. 2023 Mar 14;7(1):rkad022. doi: 10.1093/rap/rkad022. eCollection 2023. PMID 36923262
- [Background] Kowal-Bielecka O, Fransen J, Avouac J, Becker M, Kulak A, Allanore Y, Distler O, Clements P, Cutolo M, Czirjak L, Damjanov N, Del Galdo F, Denton CP, Distler JHW, Foeldvari I, Figelstone K, Frerix M, Furst DE, Guiducci S, Hunzelmann N, Khanna D, Matucci-Cerinic M, Herrick AL, van den Hoogen F, van Laar JM, Riemekasten G, Silver R, Smith V, Sulli A, Tarner I, Tyndall A, Welling J, Wigley F, Valentini G, Walker UA, Zulian F, Muller-Ladner U; EUSTAR Coauthors. Update of EULAR recommendations for the treatment of systemic sclerosis. Ann Rheum Dis. 2017 Aug;76(8):1327-1339. doi: 10.1136/annrheumdis-2016-209909. Epub 2016 Nov 9. PMID 27941129
- [Background] Khanna D, Lescoat A, Roofeh D, Bernstein EJ, Kazerooni EA, Roth MD, Martinez F, Flaherty KR, Denton CP. Systemic Sclerosis-Associated Interstitial Lung Disease: How to Incorporate Two Food and Drug Administration-Approved Therapies in Clinical Practice. Arthritis Rheumatol. 2022 Jan;74(1):13-27. doi: 10.1002/art.41933. Epub 2021 Nov 10. PMID 34313399
- [Background] Flaherty KR, Brown KK, Wells AU, Clerisme-Beaty E, Collard HR, Cottin V, Devaraj A, Inoue Y, Le Maulf F, Richeldi L, Schmidt H, Walsh S, Mezzanotte W, Schlenker-Herceg R. Design of the PF-ILD trial: a double-blind, randomised, placebo-controlled phase III trial of nintedanib in patients with progressive fibrosing interstitial lung disease. BMJ Open Respir Res. 2017 Sep 17;4(1):e000212. doi: 10.1136/bmjresp-2017-000212. eCollection 2017. PMID 29018526